CLINICAL TRIAL: NCT02544373
Title: A Randomized Trial of Positive Airway Pressure Therapy to Treat Cognitive Dysfunction in MS Patients With Obstructive Sleep Apnea
Brief Title: CPAP to Treat Cognitive Dysfunction in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Tiffany J. Braley, MD, MS, Associate Professor, Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00098738
Record Dates: First submitted 2015-05-26; First posted 2015-09-09 (Estimated); Results first posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: OSA; Obstructive Sleep Apnea; Cognition; Cognitive Dysfunction; Memory; Positive Aiway Pressure; CPAP; MS
MeSH Terms: conditions — Multiple Sclerosis; Sleep Apnea, Obstructive; Cognitive Dysfunction | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Immediate PAP therapy (Group 1) (Active Comparator): Subjects will receive PAP treatment for OSA as soon as possible after baseline PSG and repeat baseline cognitive testing 3 months after initiation of PAP therapy. PAP therapy is considered standard clinical care for OSA. It involves wearing an apparatus that includes a hose and a mask (that covers the nose, or nose and mouth), connected to a small machine that blows air into the airway during sleep. The degree of air pressure given depends on your apnea severity, and the supplied air pressure can be continuous or change with your breathing pattern (bilevel).
  Interventions: Device: PAP therapy
- Standard Care PAP therapy (Group 2) (Other): Subjects will delay PAP treatment for 3 months following their baseline sleep study, and repeat their baseline cognitive testing prior to PAP treatment for sleep apnea. PAP therapy is considered standard clinical care for OSA. It involves wearing an apparatus that includes a hose and a mask (that covers the nose, or nose and mouth), connected to a small machine that blows air into the airway during sleep. The degree of air pressure given depends on your apnea severity, and the supplied air pressure can be continuous or change with your breathing pattern (bilevel).
  Interventions: Device: PAP therapy

INTERVENTIONS:
Device: PAP therapy — Positive airway pressure treatment for obstructive sleep apnea
  Other Names: Positive airway pressure; CPAP; BiPAP; Continuous positive airway pressure; Bi-level positive airway pressure

SUMMARY:
The objectives of this study are to determine the effects of obstructive sleep apnea (OSA) on cognitive function in patients with multiple sclerosis (MS); and to evaluate whether OSA treatment with positive airway pressure therapy could improve cognitive dysfunction in MS patients who have OSA.

DETAILED DESCRIPTION:
Up to 70% of patients with MS suffer from cognitive dysfunction (difficulties with thinking, information processing, verbal expression, or memory). Cognitive dysfunction is one of the most disabling symptoms of MS, that can profoundly affect job performance, family responsibilities, and quality of life. While no treatments have been shown to improve cognitive dysfunction in MS, many patients have not been evaluated or treated for other common health problems that could be contributing to their cognitive dysfunction.

Up to 50% of MS patients also suffer from obstructive sleep apnea (OSA). Obstructive sleep apnea is a common disorder in which the upper airway collapses during sleep, causing poor sleep quality and decreased oxygen levels in the blood. In patients without MS, OSA is a well-established cause of poor cognitive performance. Recent studies of non-MS patients also suggest that cognitive performance may improve with OSA treatment. Yet, despite the high number of MS patients with OSA, the relationship between OSA and cognitive performance, and the effects of OSA treatment on cognitive performance in MS, has not received sufficient study.

The objectives of this study are to determine the effects of obstructive sleep apnea (OSA) on cognitive function in patients with multiple sclerosis (MS); and to evaluate whether OSA treatment with positive airway pressure therapy could improve cognitive dysfunction in MS patients who also have OSA.

Interested participants with MS who screen positive on a commonly used screening tool used to detect those at high risk for OSA will be invited to participate. Consenting participants will have a baseline cognitive (memory and thinking) test to assess their cognitive function, and an overnight sleep study (polysomnogram, or PSG) to determine if they have obstructive sleep apnea. If the sleep study shows signs of sleep apnea, participants will be assigned treatment for their sleep apnea with positive airway pressure (PAP) therapy, either immediately (Group 1), or 3 months after the baseline sleep study (Group 2). Groups will be assigned at random (like flipping a coin). There is a 2/3 chance that participants will be assigned to Group 1. PAP therapy is considered standard clinical care for OSA. It involves wearing an apparatus that includes a hose and a mask (that covers the nose, or nose and mouth), connected to a small machine that blows air into the airway during sleep. In order to determine which airway pressure most effectively treats an individual's sleep apnea, and what type of mask is needed, a separate sleep study known as an overnight "PAP titration study" will also be performed. This study is similar to a PSG but also involves fitting of various masks which are then hooked up to the individual and PAP machine to test the effectiveness of various PAP settings, and to determine which mask is most tolerable for the individual.

Participants will also receive repeat cognitive testing at 3 months to see if the immediate sleep apnea treatment group (Group 1) shows improvements memory and thinking, as compared to the standard care treatment group (Group 2), who will not start apnea treatment until after their repeat cognitive test. Participants will be compensated for their travel and time throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria

1. Age of 18-70 years at screening
2. Diagnosis of clinically definite MS
3. Willingness to undergo in-lab baseline polysomnography (PSG) and positive airway pressure (PAP) titration (if needed)
4. Willingness to undergo 2 separate 90-minute cognitive testing sessions
5. Either one of the following:

   Score of >=2 sleep apnea risk factors on the "STOP-Bang" sleep apnea screening questionnaire. The STOP-Bang questionnaire is a screening tool consisting of eight items which reflect OSA risk factors. STOP-Bang scores of ≥3 indicate elevated risk for moderate-severe OSA in the general population, and scores as low as 2 are frequently seen in MS patients with OSA, based on previous data from the PI).

   OR

   Have a pre-existing diagnosis of OSA based on a previous overnight sleep study (either home study or in-lab) but have not yet started using PAP therapy on a compliant basis. *If OSA was NOT diagnosed by a U-M in-lab sleep study within the past year prior to screening, subjects must be willing to get new baseline in-lab U-M PSG as part of study.
6. Willingness to start treatment with PAP if OSA present

Exclusion Criteria

1. Physical, psychiatric or cognitive impairment that prevents informed consent, PSG, PAP use, or reliable longitudinal follow-up
2. Cardiopulmonary conditions that may increase sleep apnea risk
3. Current treatment, such as PAP, for obstructive or central sleep apnea
4. History of surgical treatment for OSA
5. Nervous system diseases other than MS that may predispose subjects to OSA (such as Parkinson's disease, amyotrophic lateral sclerosis, or recent stroke)
6. History of concomitant central nervous system disease that could influence cognition, such as large vessel territory stroke, Alzheimer's disease, Parkinson's disease, or Lewy body dementia
7. Concomitant systemic autoimmune disease with secondary central nervous system involvement (including CNS lupus or neurosarcoidosis).
8. Pregnancy
9. Evidence of clinical MS relapse within the last 30 days prior to enrollment
10. Systemic high dose steroid use (1 gram IV methylprednisolone daily for 3-5 days or equivalent)for an MS relapse within the last 30 days prior to enrollment
11. Unwillingness to initiate PAP therapy if clinically indicated
12. Severe depression at screening per the Patient Health Questionnaire-8 (PHQ-8) (The PHQ-8 is a brief, self-administered questionnaire that evaluates core symptoms associated with major depressive disorder. Scores range from 0 to 24 based on the frequency and severity of depressive symptoms over the previous two weeks.)
13. Anticipated initiation, dosage change, or discontinuation in medications that could, per the opinion of the investigators, influence cognitive test scores from baseline to follow-up, including MS disease modifying therapies, hypnotic agents, narcotic-based medications, benzodiazepines, antispasmodics, or 4-aminopyridine
14. ESS scores >= 16 on baseline visit
15. Subjects with extreme OSA accompanied by signs of cardiopulmonary compromise (RDI>60 respiratory events per hour with severe nocturnal hypoxia or unstable ECG rhythms on PSG), will be excluded unless they are randomized to immediate PAP arm
16. Any other condition or treatment that in the opinion of the investigator could affect subject safety or study eligibility

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Braley, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Brassington JC, Marsh NV. Neuropsychological aspects of multiple sclerosis. Neuropsychol Rev. 1998 Jun;8(2):43-77. doi: 10.1023/a:1025621700003. PMID 9658410
- [Background] Diamond BJ, DeLuca J, Kim H, Kelley SM. The question of disproportionate impairments in visual and auditory information processing in multiple sclerosis. J Clin Exp Neuropsychol. 1997 Feb;19(1):34-42. doi: 10.1080/01688639708403834. PMID 9071639
- [Background] DeLuca J, Barbieri-Berger S, Johnson SK. The nature of memory impairments in multiple sclerosis: acquisition versus retrieval. J Clin Exp Neuropsychol. 1994 Apr;16(2):183-9. doi: 10.1080/01688639408402629. PMID 8021305
- [Background] Kujala P, Portin R, Ruutiainen J. Memory deficits and early cognitive deterioration in MS. Acta Neurol Scand. 1996 May;93(5):329-35. doi: 10.1111/j.1600-0404.1996.tb00005.x. PMID 8800343
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Background] Peyser JM, Rao SM, LaRocca NG, Kaplan E. Guidelines for neuropsychological research in multiple sclerosis. Arch Neurol. 1990 Jan;47(1):94-7. doi: 10.1001/archneur.1990.00530010120030. PMID 2403789
- [Background] Beatty WW, Paul RH, Wilbanks SL, Hames KA, Blanco CR, Goodkin DE. Identifying multiple sclerosis patients with mild or global cognitive impairment using the Screening Examination for Cognitive Impairment (SEFCI). Neurology. 1995 Apr;45(4):718-23. doi: 10.1212/wnl.45.4.718. PMID 7723961
- [Background] Knight RG, Devereux RC, Godfrey HP. Psychosocial consequences of caring for a spouse with multiple sclerosis. J Clin Exp Neuropsychol. 1997 Feb;19(1):7-19. doi: 10.1080/01688639708403832. PMID 9071637
- [Background] Rao SM, Leo GJ, Ellington L, Nauertz T, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991 May;41(5):692-6. doi: 10.1212/wnl.41.5.692. PMID 1823781
- [Background] O'Brien AR, Chiaravalloti N, Goverover Y, Deluca J. Evidenced-based cognitive rehabilitation for persons with multiple sclerosis: a review of the literature. Arch Phys Med Rehabil. 2008 Apr;89(4):761-9. doi: 10.1016/j.apmr.2007.10.019. PMID 18374010
- [Background] Canessa N, Castronovo V, Cappa SF, Aloia MS, Marelli S, Falini A, Alemanno F, Ferini-Strambi L. Obstructive sleep apnea: brain structural changes and neurocognitive function before and after treatment. Am J Respir Crit Care Med. 2011 May 15;183(10):1419-26. doi: 10.1164/rccm.201005-0693OC. Epub 2010 Oct 29. PMID 21037021
- [Background] Benedict RH, Cookfair D, Gavett R, Gunther M, Munschauer F, Garg N, Weinstock-Guttman B. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc. 2006 Jul;12(4):549-58. doi: 10.1017/s1355617706060723. PMID 16981607
- [Background] Benedict RH, Fischer JS, Archibald CJ, Arnett PA, Beatty WW, Bobholz J, Chelune GJ, Fisk JD, Langdon DW, Caruso L, Foley F, LaRocca NG, Vowels L, Weinstein A, DeLuca J, Rao SM, Munschauer F. Minimal neuropsychological assessment of MS patients: a consensus approach. Clin Neuropsychol. 2002 Aug;16(3):381-97. doi: 10.1076/clin.16.3.381.13859. PMID 12607150
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Chung F, Subramanyam R, Liao P, Sasaki E, Shapiro C, Sun Y. High STOP-Bang score indicates a high probability of obstructive sleep apnoea. Br J Anaesth. 2012 May;108(5):768-75. doi: 10.1093/bja/aes022. Epub 2012 Mar 8. PMID 22401881
- [Background] Chervin RD, Malhotra RK, Burns JW. Respiratory cycle-related EEG changes during sleep reflect esophageal pressures. Sleep. 2008 Dec;31(12):1713-20. doi: 10.1093/sleep/31.12.1713. PMID 19090327
- [Background] Chervin RD, Shelgikar AV, Burns JW. Respiratory cycle-related EEG changes: response to CPAP. Sleep. 2012 Feb 1;35(2):203-9. doi: 10.5665/sleep.1622. PMID 22294810
- [Background] Braley TJ, Segal BM, Chervin RD. Obstructive sleep apnea and fatigue in patients with multiple sclerosis. J Clin Sleep Med. 2014 Feb 15;10(2):155-62. doi: 10.5664/jcsm.3442. PMID 24532998
- [Background] Brass SD, Li CS, Auerbach S. The underdiagnosis of sleep disorders in patients with multiple sclerosis. J Clin Sleep Med. 2014 Sep 15;10(9):1025-31. doi: 10.5664/jcsm.4044. PMID 25142763
- [Background] Castronovo V, Canessa N, Strambi LF, Aloia MS, Consonni M, Marelli S, Iadanza A, Bruschi A, Falini A, Cappa SF. Brain activation changes before and after PAP treatment in obstructive sleep apnea. Sleep. 2009 Sep;32(9):1161-72. doi: 10.1093/sleep/32.9.1161. PMID 19750921
- [Background] Castronovo V, Scifo P, Castellano A, Aloia MS, Iadanza A, Marelli S, Cappa SF, Strambi LF, Falini A. White matter integrity in obstructive sleep apnea before and after treatment. Sleep. 2014 Sep 1;37(9):1465-75. doi: 10.5665/sleep.3994. PMID 25142557
- [Background] Aloia MS, Arnedt JT, Davis JD, Riggs RL, Byrd D. Neuropsychological sequelae of obstructive sleep apnea-hypopnea syndrome: a critical review. J Int Neuropsychol Soc. 2004 Sep;10(5):772-85. doi: 10.1017/S1355617704105134. PMID 15327723
- [Background] Cohen-Zion M, Stepnowsky C, Marler, Shochat T, Kripke DF, Ancoli-Israel S. Changes in cognitive function associated with sleep disordered breathing in older people. J Am Geriatr Soc. 2001 Dec;49(12):1622-7. doi: 10.1046/j.1532-5415.2001.t01-1-49270.x. PMID 11843994
- [Background] Bucks RS, Olaithe M, Eastwood P. Neurocognitive function in obstructive sleep apnoea: a meta-review. Respirology. 2013 Jan;18(1):61-70. doi: 10.1111/j.1440-1843.2012.02255.x. PMID 22913604
- [Derived] Valentine TR, Kratz AL, Kaplish N, Chervin RD, Braley TJ. Sleep-disordered breathing and neurocognitive function in multiple sclerosis: Differential associations across cognitive domains. Mult Scler. 2023 Jun;29(7):832-845. doi: 10.1177/13524585231169465. Epub 2023 May 17. PMID 37194432

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 135 enrolled participants,131 received both baseline cognitive testing and polysomnography for Aim 1 (pre-intervention) analyses (outside of the interventional phase of the study. Among these 131 participants, 111 were randomized for this trial.
Period: Overall Study
Arm/Group | Immediate PAP Therapy (Group 1) | Standard Care PAP Therapy (Group 2)
Started | 71 | 40
Completed | 58 | 35
Not Completed | 13 | 5
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data is provided for all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate PAP Therapy (Group 1) | Standard Care PAP Therapy (Group 2) | Total
Number analyzed (Participants) | 71 | 40 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9) | 49.2 (9.2) | 49.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 28 | 78
  Male | 21 | 12 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 33 | 94
  Black | 8 | 5 | 13
  Asian | 1 | 0 | 1
  American Indian/Alaskan Native | 1 | 0 | 1
  Unknown/Not reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 2 | 3
  Non-Hispanic | 69 | 37 | 106
  Unknown/Not reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 40 | 111
Apnea Hypopnea Index [Mean (Standard Deviation); unit: units on a scale] — For an Apnea-Hypopnea Index from 5 to <15 denotes mild sleep apnea. 15 to <30 is moderate, while an AHI of 30 or greater is considered severe. AHI = sum of the number of apneas (pauses in breathing) plus the number of hypopneas (periods of shallow breathing) occurring, on average, per hour of sleep.
  units on a scale | 23.1113 (19.22115) | 20.4875 (16.30875) | 22.1658 (18.19362)

OUTCOME MEASURES:

1. Primary Outcome: Association Between Obstructive Sleep Apnea (OSA) Severity [as Measured by Apnea Hypopnea Index (AHI) e.g., Number of Apneic Events Per Hour of Sleep] and Baseline Performance on the Minimal Assessment of Cognitive Function in MS Battery (MACFIMS)
Description: Bivariate associations between AHI measured with PSG, and baseline MACFIMS test results which include:
  * Controlled Oral Word Association Test (COWAT): verbal fluency;
  * Judgement of Line Orientation test (JLO): visuospatial perception;
  * Brief Visuospatial Memory Test Revised Total (BVMT-R Total) and Brief Visuospatial Memory Test Revised Delayed (BVMT-R Delayed): visual memory & learning;
  * California Verbal Learning Test-II Total score (CVLT-II): verbal memory & learning;
  * Paced Auditory Serial Addition Test-2 (PASAT-2), Paced Auditory Serial Addition Test-3 (PASAT-3) and Symbol Digit Modalities test (SDMT): memory, attention, processing speed.
  For each test higher scores indicate better cognitive performance. Beta coefficients were generated with multiple linear regression models, yielding the confidence intervals shown below.
Time Frame: Participants had up to 3 weeks to complete both baseline cognitive testing and PSG
Population: These analyses were conducted to examine associations between apnea severity and cognitive performance prior to randomization and PAP intervention. Four out of 135 consented had missing data that did not allow analysis of associations.
Measure: Number (95% Confidence Interval); unit: beta coefficient
Groups:
- All Participants Prior to Randomization: All participants who received both baseline cognitive testing and diagnostic polysomnography (PSG), prior to randomization. Participants who did not have obstructive sleep apnea (OSA) on PSG concluded the study prior to randomization.
Arm/Group | All Participants Prior to Randomization
Number analyzed (Participants) | 131
beta coefficient
  COWAT | -0.014 [-0.126 to 0.099]
  JLO | -0.003 [-0.044 to 0.037]
  BVMT-R Total | -0.061 [-0.124 to 0.001]
  BVMT-R Delayed | -0.026 [-0.051 to -0.001]
  CVLT-II Total | 0.009 [-0.117 to 0.135]
  PASAT-2 Total | -0.022 [-0.130 to 0.086]
  PASAT-3 Total | -0.061 [-0.189 to 0.067]
  SDMT | -0.137 [-0.268 to -0.007]

2. Primary Outcome: Change From Baseline in Performance on the Minimal Assessment of Cognitive Function in MS Battery (MACFIMS)
Description: Mean change in scores on individual MACFIMS tests from baseline to month 3 cognitive testing, as calculated by Month 3 minus baseline score shown by treatment group. MACFIMS tests with score ranges (minimum-maximum) are listed here:
  * Controlled Oral Word Association Test (COWAT) 0 - no recognized upper limit;
  * Judgement of Line Orientation test (JLO) 0-34 based on scores adjusted for age and sex;
  * Brief Visuospatial Memory Test Revised Total (BVMT-R Total) 0-36;
  * Brief Visuospatial Memory Test Revised Delayed (BVMT-R Delayed), 0-12;
  * California Verbal Learning Test-II Total score (CVLT-II); (T scores necessary for analysis; 50=population mean; 10=SD);
  * Paced Auditory Serial Addition Test-2 (PASAT-2), 0-60;
  * Paced Auditory Serial Addition Test-3 (PASAT-3) 0-60; and
  * Symbol Digit Modalities test (SDMT) 0-110. For all measures, higher scores mean better performance, so based on subtracting 3 month values minus baseline, any positive numbers indicate improvement.
Time Frame: baseline, 3 months
Population: includes participants who had MACFIMS testing at both timepoints (baseline and month 3)
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Immediate PAP Therapy (Group 1) | Standard Care PAP Therapy (Group 2)
Number analyzed (Participants) | 71 | 40
score
  COWAT | 2.5 (8.23) | 2.69 (8.35)
  JLO | 0.28 (2.78) | 0.60 (3.39)
  BVMT-R Total | 1.81 (5.04) | 1.43 (4.99)
  BVMT-R Delayed | 0.95 (1.99) | 0.54 (1.88)
  CVLT-II | 2.84 (9.59) | 4.77 (8.88)
  PASAT-2 | 2.27 (6.95) | 2.09 (5.14)
  PASAT-3 | 0.61 (7.16) | 2.53 (8.33)
  SDMT | 0.16 (6.24) | 1.03 (6.72)

3. Other Pre Specified Outcome: Association Between Polysomnographic Measures of Sleep Efficiency (Ratio of Time Spent Asleep to Total Time in Bed) and Baseline Performance on the Minimal Assessment of Cognitive Function in MS Battery (MACFIMS)
Time Frame: 3 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Association Between Wake Time After Sleep Onset (Total Time in Minutes Spent Awake After Sleep Onset, and Before Final Awakening Time) and Baseline Performance on the Minimal Assessment of Cognitive Function in MS Battery (MACFIMS)
Time Frame: 3 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Association Between the Total Arousal Index (Average Number of EEG Arousals Per Hour of Sleep) and Baseline Performance on the Minimal Assessment of Cognitive Function in MS Battery (MACFIMS)
Time Frame: 3 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Association Between Sleep Stage Percentages (% Total Sleep Time Spent in Stage N1, N2, N3, and REM Sleep) and Baseline Performance on the Minimal Assessment of Cognitive Function in MS Battery (MACFIMS)
Time Frame: 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE data were collected from the time participants were randomized until 30 days after the treatment period (per protocol = 3 month treatment period + 30 day post-treatment = 4 months).
Arm/Group | Immediate PAP Therapy (Group 1) | Standard Care PAP Therapy (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/40
Other Adverse Events (participants affected / at risk) | 11/71 | 0/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate PAP Therapy (Group 1) (N=71) | Standard Care PAP Therapy (Group 2) (N=40)
Common cold (Infections and infestations) | 6 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT02544373/Prot_SAP_000.pdf